CLINICAL TRIAL: NCT00906880
Title: Clinical Study to Assess the Clinical Tolerability, Feasibility and Effectiveness Under Field Conditions of the Combination of Nifurtimox and Eflornithine (NECT) for the Treatment of T.b.Gambiense Human African Trypanosomiasis (HAT) in the Meningo-encephalitic Stage
Brief Title: Clinical Study to Assess the Tolerability, Feasibility and Effectiveness of Nifurtimox and Eflornithine (NECT) for the Treatment of Trypanosoma Brucei Gambiense Human African Trypanosomiasis (HAT) in the Meningo-encephalitic Phase
Acronym: NECT-FIELD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAT0208
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Human African Trypanosomiasis
Keywords: Human African Trypanosomiasis; HAT; sleeping sickness; combination treatment; nifurtimox; eflornithine; Human African Trypanosomiasis in the meningo-encephalitic phase (stage 2 HAT)
MeSH Terms: conditions — Trypanosomiasis, African | interventions — Nifurtimox; Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nifurtimox-Eflronithine Combination Treatment (NECT) — co-administration of nifurtimox (10 days, 15 mg/kg/day, p.o. TID) and eflornithine (7 days, 400 mg/kg/day, i.v. BID)
  Other Names: nifurtimox (Lampit); eflornithine (Ornidyl)

SUMMARY:
Multicenter, open label, uncontrolled phase IIIb study of therapeutic use of the combination of nifurtimox and eflornithine (NECT) for the treatment of Trypanosoma brucei gambiense human African trypanosomiasis (HAT) in the meningo-encephalitic phase.

Overall objectives:

Assess the clinical tolerability, feasibility and effectiveness of NECT co-administration to treat patients with T.b. gambiense human African trypanosomiasis (HAT) in the meningo-encephalitic phase in actual real-life conditions (regular treatment centers of the National HAT Control Programme, NGO treatment centers).

Primary objective:

* Assess the clinical response of the NECT co-administration under field conditions.

Secondary objectives:

* Assess the incidence and type of adverse events (AE), and the capacity of the treatment centers to deal with these.
* Assess the feasibility of the implementation of the NECT coadministration by the health center.
* Assess the effectiveness of the NECT co-administration at 24* months after treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed as stage 2 HAT according to the diagnostic protocols in use at the treatment center (generally, if presence of parasites in blood, lymph node fluid or CSF and an elevated white blood cell count in the CSF, but this can vary from center to center) will be included if a written Informed Consent is given by the patient or a legally acceptable representative if the patient is a minor or unable to communicate.

* Pregnancy and breastfeeding women: On a case by case basis according to the guidelines of the National HAT Control Programme or the NGO, the Investigator will decide to treat the patient or to defer the treatment. In case of inclusion, the mother-child pairs or the children of lactating mothers will be closely monitored during treatment and follow up.
* Children under 2 years of age: On a case by case basis, the Investigator will decide to treat an infant with NECT or an alternative treatment (preferably eflornithine). In case of inclusion, these infants will be closely monitored during treatment and follow up like all children less than 12 years of age.

Exclusion Criteria:

* Unable to take oral medication, and impossibility to use a nasogastric tube.
* Treatment failure after nifurtimox-eflornithine treatment.
* Any other condition or reason for which the Investigator (or the responsible treating staff member) judges that another or no HAT treatment is warranted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients discharged alive from the hospital or the treatment center

SECONDARY OUTCOMES:
Incidence of serious AE (SAE) and severe AE (CTC score 3 and 4) related to treatment, and overall frequency and nature of AE and need for additional medications to manage these. | up to 24 months after treatment
Effectiveness: The clinical cure rate (Survival without clinical and/or parasitological signs of HAT) | 24 months after treatment
Number of temporary treatment interruptions, number of premature treatment cessations, length of hospitalization stay (including observation period), treatment compliance (deviation in dosing), and other feasibility indicators. | during the treatment/hospitalisation time

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Blum, MD, Principal Investigator — Swiss Tropical & Public Health Institute; Victor Kande, MD, Principal Investigator — PNLTHA-DRC;
Locations (6):
- Republic of the Congo (6):
  - HGR (General Reference Hospital) Bandundu, Bandundu, Bandundu
  - HGR (General Reference Hospital) Kwamouth, Kwamouth, Bandundu
  - HGR (General Reference Hospital) Yasa Bonga, Yasa Bonga, Bandundu
  - CDTC (Centre de Dépistage, Traitement et Contrôle) Katanda, Katanda, East Kasai
  - CRT (Centre de Réference et de Traitement) Dipumba, Dipumba general hospital, Mbuji Mayi, East Kasai
  - HGR (General Reference Hospital) Ngandajika, Ngandajika, East Kasai

REFERENCES:
- [Result] Schmid C, Kuemmerle A, Blum J, Ghabri S, Kande V, Mutombo W, Ilunga M, Lumpungu I, Mutanda S, Nganzobo P, Tete D, Mubwa N, Kisala M, Blesson S, Mordt OV. In-hospital safety in field conditions of nifurtimox eflornithine combination therapy (NECT) for T. b. gambiense sleeping sickness. PLoS Negl Trop Dis. 2012;6(11):e1920. doi: 10.1371/journal.pntd.0001920. Epub 2012 Nov 29. PMID 23209861
- [Derived] Kuemmerle A, Schmid C, Bernhard S, Kande V, Mutombo W, Ilunga M, Lumpungu I, Mutanda S, Nganzobo P, Tete DN, Kisala M, Burri C, Blesson S, Valverde Mordt O. Effectiveness of Nifurtimox Eflornithine Combination Therapy (NECT) in T. b. gambiense second stage sleeping sickness patients in the Democratic Republic of Congo: Report from a field study. PLoS Negl Trop Dis. 2021 Nov 8;15(11):e0009903. doi: 10.1371/journal.pntd.0009903. eCollection 2021 Nov. PMID 34748572
- [Derived] Kuemmerle A, Schmid C, Kande V, Mutombo W, Ilunga M, Lumpungu I, Mutanda S, Nganzobo P, Ngolo D, Kisala M, Valverde Mordt O. Prescription of concomitant medications in patients treated with Nifurtimox Eflornithine Combination Therapy (NECT) for T.b. gambiense second stage sleeping sickness in the Democratic Republic of the Congo. PLoS Negl Trop Dis. 2020 Jan 27;14(1):e0008028. doi: 10.1371/journal.pntd.0008028. eCollection 2020 Jan. PMID 31986140
- See also: Sponsor website — http://www.dndi.org/